CLINICAL TRIAL: NCT04568850
Title: Waxing and Waning of Serum SARS CoV 2 IgG Level: A Prospective Study
Brief Title: Waxing and Waning of Serum SARS CoV-2-IgG Level in COVID-19 Exposed Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Amina Asif, Assistant Professor, Lahore General Hospital
Other Study IDs: LGH007
Record Dates: First submitted 2020-09-21; First posted 2020-09-29 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma of the subjects will be saved,
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Plasma IgG levels — Plasma IgG levels of subjects who tested reactive for IgG SARS CoV-2 antibodies will be monitored every month for 4 months for IgG levels

SUMMARY:
This study will define the kinetics of IgG responses to both N and S proteins in the subjects who suffered from COVID 19 and then had recovered and those who were previously undiagnosed but were seropositive. These subjects will be followed for four months to evaluate the levels of antibodies in these people.

DETAILED DESCRIPTION:
Since December 2019, cases of unexplained pneumonia have occurred in Wuhan City, Hubei Province, subsequent virus isolation and whole-genome sequencing (accession#: MN908947) confirmed that it is an acute respiratory infection caused by new severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) . Coronaviruses are enveloped, non-segmented, single-positive-stranded RNA viruses with round or oval particles and a diameter of 50-200 nm. Coronavirus subfamily is divided into four genera: α, β, γ and δ according to serotype and genomic characteristics. The SARS-CoV-2 belongs to the genus β which has been confirmed to be highly infectious by research.

The four major structural proteins of coronavirus are the spike surface glycoprotein (S), small envelope protein (E), matrix protein (M), and nucleocapsid protein (N). The spike protein (S) of coronavirus is a type I transmembrane glycoprotein and mediates the entrance to human respiratory epithelial cells by interacting with cell surface receptor angiotensin-converting enzyme 2 (ACE2), the S protein contains distinct functional domains near the amino (S1) and carboxy (S2) termini, the peripheral S1 portion can independently bind cellular receptors while the integral membrane S2 portion is required to mediate fusion of viral and cellular membranes . The nucleocapsid protein (N) forms complexes with genomic RNA, interacts with the viral membrane protein during virion assembly and plays a critical role in enhancing the efficiency of virus transcription and assembly The seropositivity rate of both IgM and IgG responses after onset and recovery of disease, and in the context of both N protein and S protein has not been clarified. The kinetics of antibody responses in critical cases or ICU patients has not been reported, and no studies have suggested whether antibody response is associated with disease prognosis

ELIGIBILITY:
Inclusion Criteria:

* Subjects testing reactive for SARS CoV 2 IgG antibodies

Exclusion Criteria:

* Subjects testing nonreactive for SARS CoV-2 IgG antibodies

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: subjects who suffered from COVID 19 and then had recovered and those who were previously undiagnosed but were seropositive.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Serum IgG for SARS CoV 2 will be monitored | 5 months
  Subjects testing reactive for SARS CoV 2 IgG antibodies will be followed for five months to see the levels of IgG SARS CoV 2

CONTACTS AND LOCATIONS:
Overall Officials: Amina Asif, MPhilMicro, Principal Investigator — Lahore General Hospital
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided